CLINICAL TRIAL: NCT02714452
Title: A Person-centred and Thriving Promoting Care Model for Residential Aged Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University of Oslo (Other); La Trobe University (Other)
Responsible Party: Principal Investigator, David Edvardsson, Professor, Umeå University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-4016
Record Dates: First submitted 2016-03-07; First posted 2016-03-21 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Aging
Keywords: Person-centred care; Thriving; Satisfaction with care; Residential aged care; Caring environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Other): Person-centred care
  Interventions: Behavioral: Person-centred care
- Control (No Intervention): Conventional care

INTERVENTIONS:
Behavioral: Person-centred care — Person-centred and thriving promoting care
  Arms: Intervention

SUMMARY:
The overall aim of this study is to evaluate the effects, meaning and significance of a person-centred and thriving promoting model for residential aged care in Australia, Norway and Sweden. More specifically, the following research questions will be explored:

1. Can a person-centred and thriving promoting care model increase residents' thriving, and have a positive impact on residents' perception of the caring environment?
2. Can a person-centred and thriving promoting care model increase relatives' satisfaction with care, and have a positive impact on their experience of visiting their relative, and perception of the caring environment?
3. Can a person-centred and thriving promoting care model increase staff's job satisfaction, decrease stress of conscience, and have a positive impact on their perception of the caring environment and person-centred care?
4. What meaning and significance do relatives and staff ascribe to the intervention? The study is designed as a multi-centre, controlled group before-after design with participating sites in Victoria (Australia), Oslo (Norway) and Västerbotten (Sweden). Two residential aged care facilities at each site will be allocated to either intervention or control, in total three intervention and three control facilities divided over the three sites.

Care staff at the intervention facilities will participate in a 12-month education on how to integrate aspects of person-centredness, thriving and a caring environment into daily care practice. Participating staff will work together with their colleagues and members from the research group to create a reflective and creative learning environment that builds on and develops the staff members' clinical experience and skills, and combines it with theoretical and research-based knowledge.

At the control facilities, care staff will participate in a 2-hour lecture on the theoretical and philosophical foundations of person-centredness, thriving and a caring environment, and then continue with practice without further involvement from the research team.

Evaluation data will be collected by study specific questionnaires before the education starts, immediately after the education and at a 6-month follow-up. In addition, focus group interviews and individual interviews will be conducted with a selection of staff members and relatives at the intervention facilities to explore meaning and significance of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years of age
* living in the facility for >1 month by the time of data collection
* visiting the residential aged care facility on a regular basis (>1/month)
* working in the residential aged care facility on a temporary and or permanent basis (>1month contract)
* have been working >1 month in the residential aged care facility by the time of data collection.

Exclusion Criteria:

* newly moved in to the facility
* visiting the facility more seldom than once a month
* working on a short-term contract

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in The Thriving of Older People Assessment Scale between baseline and follow-up | Change from baseline thriving at 12 and 18 months
  Data will be collected from residents at both intervention and control facilities by either self-rating or proxy-rating surveys at baseline and at 12 and 18 months follow-up
Change in relatives' satisfaction with care measured by the Pyramid questionnaire | Change from baseline satisfaction at 12 and 18 months
  Data will be collected from relatives at both intervention and control facilities by self-rating surveys at baseline and at 12 and 18 months follow-up
Change in staff's job satisfaction measured by the The Job satisfaction questionnaire | Change from baseline job satisfaction at 12 and 18 months
  Data will be collected from staff at both intervention and control facilities by self-rating surveys at baseline and at 12 and 18 months follow-up

SECONDARY OUTCOMES:
Change in participants' experience of the caring environment measured by The Person-centred Climate Questionnaire | Change from baseline experience at 12 and 18 months
  Data will be collected from residents, relatives and staff at both intervention and control facilities by either self-rating or proxy-rating surveys at baseline and at 12 and 18 months follow-up
Change in relatives' experienced satisfaction with visiting the nursing home and their relative, measured by Visual Analogue Scales of participants' subjective experiences of 12 statements, ranging from 0 (totally disagree) to 10 (totally agree). | Change from baseline satisfaction at 12 and 18 months
  Data will be collected from relatives at both intervention and control facilities by self-rating surveys at baseline and at 12 and 18 months follow-up. Group level data will be aggregated using mean values of the participants' ratings.
Change in staff's stress of conscience measured by the Stress of Conscience questionnaire | Change from baseline stress of conscience at 12 and 18 months
  Data will be collected from staff at both intervention and control facilities by self-rating surveys at baseline and at 12 and 18 months follow-up
Change in staff's perception of the person-centredness of care measured by the Person-centred Care Assessment Tool | Change from baseline perception at 12 and 18 months
  Data will be collected from staff at both intervention and control facilities by self-rating surveys at baseline and at 12 and 18 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David Edvardsson, Professor, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sjogren K, Bergland A, Kirkevold M, Lindkvist M, Lood Q, Sandman PO, Vassbo TK, Edvardsson D. Effects of a person-centred and thriving-promoting intervention on nursing home residents' experiences of thriving and person-centredness of the environment. Nurs Open. 2022 Jul;9(4):2117-2129. doi: 10.1002/nop2.1222. Epub 2022 Apr 29. PMID 35485234
- [Derived] Vassbo TK, Bergland A, Kirkevold M, Lindkvist M, Lood Q, Sandman PO, Sjogren K, Edvardsson D. Effects of a person-centred and thriving-promoting intervention on nursing home staff job satisfaction: A multi-centre, non-equivalent controlled before-after study. Nurs Open. 2020 Jul 23;7(6):1787-1797. doi: 10.1002/nop2.565. eCollection 2020 Nov. PMID 33072363
- [Derived] Lood Q, Sjogren K, Bergland A, Lindkvist M, Kirkevold M, Sandman PO, Edvardsson D. Effects of a staff education programme about person-centred care and promotion of thriving on relatives' satisfaction with quality of care in nursing homes: a multi-centre, non-equivalent controlled before-after trial. BMC Geriatr. 2020 Aug 1;20(1):268. doi: 10.1186/s12877-020-01677-7. PMID 32738880
- [Derived] Edvardsson D, Sjogren K, Lood Q, Bergland A, Kirkevold M, Sandman PO. A person-centred and thriving-promoting intervention in nursing homes - study protocol for the U-Age nursing home multi-centre, non-equivalent controlled group before-after trial. BMC Geriatr. 2017 Jan 17;17(1):22. doi: 10.1186/s12877-016-0404-1. PMID 28095791